CLINICAL TRIAL: NCT00513695
Title: A Phase II Study Evaluating the Safety and Efficacy of Sunitinib Maleate in Combination With Weekly Paclitaxel Followed by Doxorubicin and Daily Oral Cyclophosphamide Plus G-CSF as Neoadjuvant Chemotherapy for Locally Advanced or Inflammatory Breast Cancer
Brief Title: Sunitinib Malate, Paclitaxel, Doxorubicin Hydrochloride, and Cyclophosphamide Before Surgery in Treating Patients With Stage IIB-IIIC Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Specht, Principal Investigator, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6488; NCI-2010-00607 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCT00831584 (obsolete NCT alias)
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Inflammatory Breast Cancer; Male Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Inflammatory Breast Neoplasms; Breast Neoplasms, Male; Breast Neoplasms | interventions — Sunitinib; Paclitaxel; Taxes; Doxorubicin; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (neoadjuvant chemotherapy before surgery) (Experimental): Patients receive neoadjuvant chemotherapy comprising sunitinib malate PO once daily and paclitaxel IV over 1 hour once weekly for 8-12 weeks in the absence of disease progression or unacceptable toxicity. Beginning within 3 weeks of completion of sunitinib malate and paclitaxel, patients receive doxorubicin IV once weekly for 15 weeks, cyclophosphamide PO once daily for 15 weeks, and filgrastim SC on days 2-7 for 16 weeks in the absence of disease progression or unacceptable toxicity. Beginning 3-6 weeks after completion of chemotherapy, patients undergo surgery.
  Interventions: Drug: sunitinib malate; Drug: paclitaxel; Drug: doxorubicin hydrochloride; Drug: cyclophosphamide; Biological: filgrastim; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Other: flow cytometry

INTERVENTIONS:
Drug: sunitinib malate — Given PO
  Other Names: SU11248; sunitinib; Sutent
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: cyclophosphamide — Given PO
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Procedure: therapeutic conventional surgery — Undergo surgery
Other: laboratory biomarker analysis — Correlative studies
Other: flow cytometry — Correlative studies

SUMMARY:
This phase II trial studies how well giving sunitinib malate together with paclitaxel, doxorubicin hydrochloride, and cyclophosphamide before surgery works in treating patients with stage IIB-IIIC breast cancer. Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor. Drugs used in chemotherapy, such as paclitaxel, doxorubicin hydrochloride, and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sunitinib malate together with combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I.To assess the microscopic pathologic complete response rate (pCR) in patients treated with a two part, neoadjuvant regimen consisting of daily oral sunitinib with weekly IV paclitaxel for 12 weeks followed by weekly doxorubicin and daily oral cyclophosphamide given with filgrastim (G-CSF) support for 15 weeks.

SECONDARY OBJECTIVES:

I. To assess the association between microscopic pCR and clinical complete response rate at the primary tumor site.

II. To assess the relapse rate, overall and disease-free survival in patients with breast cancer treated with neoadjuvant chemotherapy consisting of daily oral sunitinib with weekly IV paclitaxel for 12 weeks followed weekly doxorubicin and daily oral cyclophosphamide given with G-CSF support for 15 weeks.

III. To assess the toxicity associated with these regimens. IV. To explore the relationship between planned correlative laboratory and clinical studies and indicators of efficacy such as pathologic response, clinical response and relapse.

OUTLINE:

Patients receive neoadjuvant chemotherapy comprising sunitinib malate orally (PO) once daily and paclitaxel intravenously (IV) over 1 hour once weekly for 8-12 weeks in the absence of disease progression or unacceptable toxicity. Beginning within 3 weeks of completion of sunitinib malate and paclitaxel, patients receive doxorubicin IV once weekly for 15 weeks, cyclophosphamide PO once daily for 15 weeks, and filgrastim subcutaneously (SC) on days 2-7 for 16 weeks in the absence of disease progression or unacceptable toxicity. Beginning 3-6 weeks after completion of chemotherapy, patients undergo surgery.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Be informed of the investigational nature of the study and all pertinent aspects of the trial and must sign and give written consent in accordance with institutional and federal guidelines
* Have a histologically-confirmed diagnosis of breast cancer that is locally advanced or inflammatory; inflammatory breast cancer is defined as erythema and peau d'orange involving half or more of the breast with a histologic diagnosis of breast cancer; the finding of focal dermal lymphatic involvement on histology does not constitute inflammatory breast cancer
* Have selected stage IIB (T3, N0, M0) or IIIA (T3, N1-2, M0 or T0-2, N2, M0) disease judged primarily unresectable by an experienced breast surgeon or otherwise deemed appropriate candidates for neoadjuvant treatment or stage IIIB (T4, any N, M0) or stage IIIC (any T, N3, M0) disease
* Patients must have a performance status of 0-2 by Zubrod criteria
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3
* Platelet count >= 100,000 cells/mm^3
* Serum creatinine =< 1.5 x institutional upper limit of normal (IULN)
* Bilirubin =< 2.0
* Serum glutamic oxaloacetic transaminase (SGOT)/serum glutamic pyruvic transaminase (SGPT)/alkaline phosphatase =< 2.0 x IULN
* Have a multi gated acquisition scan (MUGA) or echocardiogram scan performed within 3 months prior to enrollment and have a left ventricular ejection fraction (LVEF) % greater than the institutional lower limit of normal
* Be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other trial procedures

Exclusion Criteria:

* Have evidence of distant metastases
* Have tumors that overexpress human epidermal growth factor receptor 2 (HER2)/neu as evidenced by 3+ staining by immunohistochemistry or gene amplification by fluorescent in situ hybridization (FISH)
* Have received any prior chemotherapy or hormonal therapy for breast cancer
* Have received prior radiation therapy or prior definitive surgery for breast cancer
* Have a clinical diagnosis of congestive heart failure or angina pectoris or any of the following within the 6 months prior to study drug administration:, myocardial infarction, coronary/peripheral artery bypass graft, cerebrovascular accident or transient ischemic attack, or pulmonary embolism
* Have ongoing cardiac dysrhythmias of National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 3.0 grade >= 2
* Have uncontrolled hypertension (>150/100 mm Hg despite optimal medical therapy)
* Have pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
* Have a known, active infection
* Have any prior malignancy except for adequately treated basal cell or squamous cell skin cancer, any in situ cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission or any other cancer from which the patient has been disease-free for 5 years
* Human immunodeficiency virus (HIV) positive
* Are receiving or planning to receive any concurrent anticancer therapy while receiving protocol treatment
* Are receiving or planning to receive concurrent treatment on another clinical trial (supportive care trials or non-treatment trials, e.g. quality of life (QOL) are allowed; participation in the companion imaging trial, dynamic contrast enhanced-magnetic resonance imaging (DCE-MRI) and fludeoxyglucose F 18 positron emission tomography (FDG PET) with Kinetic Analysis to Monitor Breast Cancer Response to Neoadjuvant Sunitinib and Metronomic Chemotherapy is also allowed)
* Be pregnant or breast feeding; female subjects must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy; all female subjects with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment; male subjects must be surgically sterile or must agree to use effective contraception during the period of therapy; the definition of effective contraception will be based on the judgment of the principal investigator or a designated associate
* Have other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-06; Primary Completion 2012-08 (Actual); Study Completion 2017-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Specht, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (7):
- United States (7):
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Arizona Cancer Center, Tucson, Arizona
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Neoadjuvant Chemotherapy Before Surgery)
Started | 68
Completed | 63
Not Completed | 5
Not completed — Discontinued therapy | 2
Not completed — Progression prior to surgery | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Neoadjuvant Chemotherapy Before Surgery)
Number analyzed (Participants) | 68
Age, Continuous [Median (Full Range); unit: years] | 50 [33 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 50
  More than one race | 4
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Microscopic Pathologic CR (pCR) Rate
Description: Defined as no evidence of microscopic invasive tumor present at primary tumor site in the surgical specimen and calculated with exact 90% binomial confidence interval.
Time Frame: At the time of surgery
Measure: Number (95% Confidence Interval); unit: percent of evaluable participants
Arm/Group | Treatment (Neoadjuvant Chemotherapy Before Surgery)
Number analyzed (Participants) | 63
percent of evaluable participants | 27 [18 to 39]

2. Secondary Outcome: Clinical Complete Response and Correlation With Plasma VEGF, Soluble VCAM (sVCAM), and Circulating Endothelial Cells (CECs) Levels
Time Frame: At baseline, after week 12 of therapy, and prior to surgery
Population: Data not collected
Arm/Group | Treatment (Neoadjuvant Chemotherapy Before Surgery)
Number analyzed (Participants) | 0

3. Secondary Outcome: Relapse Rate
Description: Cumulative incidence rate of relapse, assessed at two years. Death is considered a competing risk.
Time Frame: Up to two years
Measure: Number (95% Confidence Interval); unit: probability of relapse
Arm/Group | Treatment (Neoadjuvant Chemotherapy Before Surgery)
Number analyzed (Participants) | 63
probability of relapse | 0.215 [0.125 to 0.322]

4. Secondary Outcome: Time to Disease Progression
Description: Median time to disease progression, at two years, as defined by clear increase in disease sites present at registration or development of new disease sites.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (Neoadjuvant Chemotherapy Before Surgery)
Number analyzed (Participants) | 63
days | NA [NA to NA] — Not reached because not enough progression events.

5. Secondary Outcome: Overall Survival
Description: Kaplan-Meier estimate from the start of protocol therapy until the date of death from any cause or the last date the patient was known to be alive, assessed at two years.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Treatment (Neoadjuvant Chemotherapy Before Surgery)
Number analyzed (Participants) | 63
survival probability | 0.875 [0.798 to 0.960]

6. Secondary Outcome: Number and Percent of Subjects Reporting Adverse Events
Description: See Adverse Events section for more details.
Time Frame: 28 days after the last dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Neoadjuvant Chemotherapy Before Surgery)
Number analyzed (Participants) | 68
Participants | 67

ADVERSE EVENTS:
Arm/Group | Treatment (Neoadjuvant Chemotherapy Before Surgery)
Serious Adverse Events (participants affected / at risk) | 47/68
Other Adverse Events (participants affected / at risk) | 67/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Neoadjuvant Chemotherapy Before Surgery) (N=68)
Neutropenia (ANC) (Blood and lymphatic system disorders) | 47
Leucopenia (Blood and lymphatic system disorders) | 23
Fatigue (General disorders) | 3
Anemia (Blood and lymphatic system disorders) | 15
Diarrhea (Gastrointestinal disorders) | 3
ALT elevation (Investigations) | 4
Rash (Skin and subcutaneous tissue disorders) | 1
Pain (General disorders) | 2
Nail changes (Skin and subcutaneous tissue disorders) | 2
Mucositis (Respiratory, thoracic and mediastinal disorders) | 7
Nausea (Gastrointestinal disorders) | 1
Sensory Neuropathy (Nervous system disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Neoadjuvant Chemotherapy Before Surgery) (N=68)
Neutropenia (ANC) (Blood and lymphatic system disorders) | 22
Leucopenia (Blood and lymphatic system disorders) | 34
Fatigue (General disorders) | 37
Anemia (Blood and lymphatic system disorders) | 32
Diarrhea (Gastrointestinal disorders) | 9
ALT elevation (Investigations) | 6
Rash (Skin and subcutaneous tissue disorders) | 8
Pain (General disorders) | 15
Hypertension (Vascular disorders) | 8
Heartburn (Gastrointestinal disorders) | 8
Nail changes (Skin and subcutaneous tissue disorders) | 12
Mucositis (Respiratory, thoracic and mediastinal disorders) | 5
Nausea (Gastrointestinal disorders) | 8
Mood alteration (Psychiatric disorders) | 7
Sensory Neuropathy (Nervous system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes